CLINICAL TRIAL: NCT00729690
Title: Effects of Oral Pregabalin on Spinal Neurotransmitters in Patients Undergoing Total Knee Replacement (TKA)
Brief Title: Effect of Oral Pregabalin on Spinal Neurotransmitters in Patients Undergoing Knee Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asokumar Buvanendran (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Asokumar Buvanendran, Attending Physician, Rush University Medical Center
Organization: Rush University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 08021105
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Results first posted 2012-12-19 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-11

CONDITIONS: PAIN
Keywords: Pregabalin; CSF; Neurotransmitter
MeSH Terms: conditions — Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 Multi-Dose Pregabalin (Experimental): Group 1 (n=16, multi-dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery and then repeat 150 mg doses at 12 and 24 hours after initial dose.
  Interventions: Drug: Pregabalin
- 2 single-dose pregabalin (Experimental): Group 2 (n=16, single dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery, and then placebo doses at 12 and 24 hours after initial dose.
  Interventions: Drug: Pregabalin
- 3 Placebo (Placebo Comparator): Group 3 (n=16, placebo): patients receive matching placebo at the same 3 time points as Groups 1 and 2.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Group 1 (n=16, multi-dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery and then repeat 150 mg doses at 12 and 24 hours after initial dose.
  Group 2 (n=16, single dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery, and then placebo doses at 12 and 24 hours after initial dose.
  Group 3 (n=16, placebo): patients receive matching placebo at the same 3 time points as Groups 1 and 2.
  Other Names: Lyrica
  Arms: 1 Multi-Dose Pregabalin
Drug: Pregabalin — Group 2 (n=16, single dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery, and then placebo doses at 12 and 24 hours after initial dose.
  Other Names: Lyrica
  Arms: 2 single-dose pregabalin
Drug: Placebo — Group 3 (n=16, placebo): patients receive matching placebo at the same 3 time points as Groups 1 and 2.
  Other Names: Lyrica
  Arms: 3 Placebo

SUMMARY:
This study involves research. Pregabalin is a Food and Drug Administration (FDA) medication approved in the United States for the treatment of nerve pain related to diabetes and post-herpetic neuralgia "shingles", and for seizures in adults. The purpose of this research is to study the effect of oral Pregabalin on spinal neurotransmitters in subjects undergoing Total Knee Replacement Surgery (TKA). TKA is associated with considerable postoperative pain which if unrelieved may result in prolonged hospital stay, inability to participate in rehabilitation programs, poor outcomes, and greater use of health-care resources. This study examines the effect of pregabalin administered for TKA on pain-related neurotransmitter concentrations.

DETAILED DESCRIPTION:
Gabapentin and the related more potent compound pregabalin have been shown to reduce postoperative pain in animal models (1). Pregabalin given before and after surgery reduced opioid use following spinal fusion surgery (2). Studies have identified the alpha 2 delta auxiliary subunit of voltage-gated calcium channels as the molecular target of pregabalin (and gabapentin), although the specific spinal site of action (presynaptic, postsynaptic) is not known.

Total knee arthroplasty (TKA) has proved to be a successful surgical treatment of knee joints affected by osteoarthritis. Currently in the United States, more than 400,000 TKAs are performed every year with reported success rates ranging from 85% to 90% (American Academy). In an aging population, the number of annual TKA procedures is expected to reach 3.48 million by the year 2030 (3).

TKA is associated with considerable postoperative pain which if unrelieved may result in prolonged hospital stay, inability to participate in rehabilitation programs, poor outcomes, and greater use of health-care resources. Perioperative pregabalin improves postoperative outcomes after TKA (4). This study examines the effect of pregabalin administered perioperatively for TKA on pain-related neurotransmitter concentrations, intrathecal analgesic consumption and range of motion (ROM). Pregabalin effects on neurotransmitter concentrations may identify pathways by which α2δ binding by pregabalin reduces postoperative pain.

Objectives:

Primary Endpoint: Measure effect of pregabalin on spinal neurotransmitters after TKA Secondary Endpoint: Correlate changes in spinal neurotransmitters with pregabalin to improvements in patient outcomes after TKA (e.g. ROM).

Other Endpoints: Suggest spinal anatomical sites of action of oral pregabalin as relates to neurotransmitter modulation and pain.

Methods:

Patient selection After approval of the Institutional Review Board of Rush University Medical Center, Chicago, Illinois, USA, 48 patients scheduled to undergo elective primary TKA by a single orthopedic surgeon will be contacted and assessed for study eligibility with a screening medical history.

A study consent form will be sent to patients who agreed to participate in the clinical study. After obtaining consent, the patient will be allocated a study number and the study drug dispensed to each participant. Using a random number table, patients will be allocated to one of three groups, without stratification by demographic characteristics:

Group 1 (n=16, multi-dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery and then repeat 150 mg doses at 12 and 24 hours after initial dose.

Group 2 (n=16, single dose pregabalin): patients receive pregabalin 150 mg orally 1 hour prior to surgery, and then placebo doses at 12 and 24 hours after initial dose.

Group 3 (n=16, placebo): patients receive matching placebo at the same 3 time points as Groups 1 and 2.

The 12 hour dosing interval was based on our pharmacokinetic study showing that after a 300 mg oral pregabalin dose, cerebrospinal fluid (CSF) pregabalin concentration reaches its peak at 8 h or later (5). Study drug administration on the day of surgery was timed to precede surgical incision by 60 +/- 30 minutes.

The physicians and nurses managing the patient during surgery and in the recovery room, the personnel involved with postoperative pain assessment and management of the intrathecal infusion, and the study patients will be blinded to group assignments. Treatment assignment codes will not be available to the investigators until all patients completed the study. A global pain score using the visual analogue scale (VAS) with 0 corresponding to "no pain" and 10 to "the worst imaginable pain" for the patient will be obtained before surgery. In the operating room, patients will be sedated with midazolam (0.05 mg/kg titrated to effect) and an intrathecal catheter placed in the sitting position, at the L3-4 or L4-5 vertebral level to deliver spinal anesthesia with bupivacaine 0.5%, (7.5 mg) and fentanyl 25mcg. Subjects will be maintained at normothermia in the operating room. A sensory analgesic level of T10 will be obtained prior to commencement of surgery. At completion of surgery an intrathecal infusion of fentanyl 0.5 mcg/ml and bupivacaine 0.1 mg/ml will be initiated using a continuous basal infusion with superimposed patient controlled intrathecal analgesia (PCIA) bolus doses. Initial infusion rates will be 4 ml/h basal intrathecal infusion plus PCIA of 1 ml q 12 min with a 4-hour lockout of 40 ml. The patients will be instructed prior to surgery to use PCIA mode at their discretion to maintain the VAS pain score <4, following a previously applied protocol (6). A standardized surgical technique will be used in all subjects.

The intrathecal catheter will be left in place for 32 h postoperatively to provide analgesia, and lumbar CSF (0.5 ml) will be withdrawn (0.5 mL) at 2, 4, 8, 12, 24, and 32 h after the initial oral dose. CSF will be frozen at -80 Centigrade (C) for subsequent assay of neurotransmitter levels. Even though CSF pregabalin does not reach its peak concentration until at least 8 h after an oral dose, earlier time points are important because:

1. Even at 2 h post-dose the CSF pregabalin concentration is already 29% of peak value, and may cause changes in neurotransmitter levels, compared to placebo.
2. CSF inflammatory mediators, such as Interleukin-6 (IL-6), increase as early as 3 h after start of surgery after total hip arthroplasty (7), and so it can be expected that neurotransmitter levels will also show early changes due to the TKA surgery alone. Any characterization of pregabalin effects on neurotransmitters after surgery needs to also measure these early changes in neurotransmitter levels, since later time points (e.g. 24 h) are not independent of events occurring earlier.

Adverse Events:

Any adverse events will be noted and reported.

ELIGIBILITY:
Inclusion Criteria:

* History of osteoarthritis
* Subjects who can understand and communicate in English

Exclusion Criteria:

* Younger than 55 years or older than 75 years.
* American Society of Anesthesiologists physical status IV
* Prior use of pregabalin or gabapentin will not be an exclusionary criterion; however patients will have been withdrawn from these medications at least 14 days before surgery
* Patients who are currently enrolled in another investigational study.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-08; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asokumar Buvanendran, MD, Principal Investigator — Rush University Medical Center; Jeffery S Kroin, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Result] Buvanendran A, Kroin JS, Della Valle CJ, Moric M, Tuman KJ. Cerebrospinal fluid neurotransmitter changes during the perioperative period in patients undergoing total knee replacement: a randomized trial. Anesth Analg. 2012 Feb;114(2):434-41. doi: 10.1213/ANE.0b013e31823dc5fb. Epub 2011 Dec 9. PMID 22156332

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-eight patients scheduled to undergo elective primary Total Knee Replacement (TKR) for osteoarthritis by 2 orthopedic surgeons were recruited at the Rush University Medical Center (Chicago, Illinois).
Groups:
- 1 Multi-Dose Pregabalin: Multi-dose pregabalin: patients receive pregabalin 150 mg orally 1 hour prior to surgery and then repeat 150 mg doses at 12 and 24 hours after initial dose.
- 2 Single-dose Pregabalin: Single dose pregabalin: patients receive pregabalin 150 mg orally 1 hour prior to surgery, and then placebo doses at 12 and 24 hours after initial dose.
- 3 Placebo: Placebo: patients receive matching placebo at the same 3 time points as Groups 1 and 2 (orally 1 hour prior to surgery and then repeat doses at 12 and 24 hours after initial dose.)
Period: Overall Study
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo
Started | 16 | 16 | 16
Completed | 16 | 14 | 14
Not Completed | 0 | 2 | 2
Not completed — IT Catheter Malfunction | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 66.9 (6.4) | 64.8 (4.4) | 66.4 (4.5) | 66.1 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 13 | 34
  Male | 4 | 7 | 3 | 14
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: NRS Pain Score AUC (NRS*hr) - 1st 24 Hours
Description: Numerical Response scale NRS(0-10) Pain scores were collected every 4 hours after the initial dose and the Area Under the Curve (AUC) calculated. Calculated for the 1st 24 hours after initial dose (0-24hr). AUC measured in NRS pain score points per hour (NRS*hr). Larger AUC values indicate higher levels of reported pain.
Time Frame: 24 hours
Population: All Completed Patients were included in the analysis.
Measure: Mean (Standard Deviation); unit: Area (NRS*hr)
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo
Number analyzed (Participants) | 16 | 14 | 14
Area (NRS*hr) | 70.4 (34.4) | 59.6 (31.1) | 73.4 (34.6)
Statistical Analysis 1: Comparison: 1 Multi-Dose Pregabalin vs 2 Single-dose Pregabalin vs 3 Placebo; For 1st 24 hours NRS AUC Pain scores; Test type: Superiority or Other; p = 0.4742, ANOVA

2. Secondary Outcome: Active Knee Flexion
Description: The degree of active knee flexion (ROM) tolerated by the patient will be assessed at days 1 and 2 post-surgery. Active flexion is the unassisted moment of the joint by the subject. On postoperative (PostOp) day 2
Time Frame: PostOp day 2
Population: All completed patients used.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo
Number analyzed (Participants) | 16 | 14 | 14
Degrees | 78.1 (10.6) | 80.5 (10.1) | 80.5 (7.0)
Statistical Analysis 1: Comparison: 1 Multi-Dose Pregabalin vs 2 Single-dose Pregabalin vs 3 Placebo; Test type: Superiority or Other; p = 0.7596, ANOVA

3. Primary Outcome: NRS Pain Score AUC (NRS*hr) - 1st 12 Hours
Description: Numerical Response scale NRS(0-10) Pain scores were collected every 4 hours after the initial dose and the Area Under the Curve (AUC) calculated. Calculated for the 1st 12 hours after initial dose (0-12hr). AUC measured in NRS pain score points per hour (NRS*hr). Larger AUC values indicate higher levels of reported pain.
Time Frame: 12 hours Post dose
Population: All Completed Patients
Measure: Mean (Standard Deviation); unit: Area (NRS*hr)
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo
Number analyzed (Participants) | 16 | 14 | 14
Area (NRS*hr) | 30.1 (15.6) | 22.7 (16.9) | 27.7 (16.7)
Statistical Analysis 1: Comparison: 1 Multi-Dose Pregabalin vs 2 Single-dose Pregabalin vs 3 Placebo; Test type: Superiority or Other; p = 0.4321, ANOVA

4. Secondary Outcome: Passive Knee Flexion
Description: Passive flexion is the moment of the joint with the assistance of a clinician (The clinician or therapist physically hold and moves the knee through it's range of motion).
Time Frame: PostOp day 2
Population: All Completed Patients were used
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo
Number analyzed (Participants) | 16 | 14 | 14
Degrees | 86.5 (15.3) | 88.2 (9.44) | 87.1 (10.6)
Statistical Analysis 1: Comparison: 1 Multi-Dose Pregabalin vs 2 Single-dose Pregabalin vs 3 Placebo; Test type: Superiority or Other; p = 0.9361, ANOVA

ADVERSE EVENTS:
Arm/Group | 1 Multi-Dose Pregabalin | 2 Single-dose Pregabalin | 3 Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 2/16 | 3/16 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Multi-Dose Pregabalin (N=16) | 2 Single-dose Pregabalin (N=16) | 3 Placebo (N=16)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No